CLINICAL TRIAL: NCT04485585
Title: An Open Label, One-sequence, 3-period Study to Evaluate Drug-drug Interactions Between BR9006-1 and BR9006-2 in Healthy Male Volunteers.
Brief Title: A Study to Evaluate Drug-drug Interactions Between BR9006-1 and BR9006-2 in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-TMC-CT-101
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Overactive Bladder
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive | interventions — Tamsulosin; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence T/M/T+M (Experimental): A total of 36 subjects will be enrolled in one sequence group. The investigational products (IPs) will be administered according to the treatment groups(T, M, T+M) assigned to on sequence group in Period 1, Period 2, and Period 3.
  * Period 1(T): BR9006-1 (Tamsulosin HCL 0.2mg) - 1 capsule QD, five-day repeated-dose
  * Period 2(M): BR9006-2 (Mirabegron 50mg) - 1 tablet QD, eleven-day repeated-dose
  * Period 3(T+M): BR9006-1 (Tamsulosin HCL 0.2mg) 1 capsule + BR9006-2 (Mirabegron 50mg) 1 tablet QD, five-day repeated-dose
  * Washout period between Period 1 and Period 2: five days
  * Washout period between Period 2 and Period 3: none
  Interventions: Drug: BR9006-1; Drug: BR9006-2

INTERVENTIONS:
Drug: BR9006-1 — * Administration to the T/T+M group: 0.2 mg of BR9006-1 will be administered one capsule once a day, five-day repeated-dose
  Other Names: Tamsulosin HCL
Drug: BR9006-2 — * Administration to the M group: 50 mg of BR9006-2 will be administered one tablet once a day, eleven-day repeated-dose
  * Administration to the T+M group: 50 mg of BR9006-2 will be administered one tablet once a day, five-day repeated-dose
  Other Names: Mirabegron

SUMMARY:
To evaluate the influence of BR9006-1 and BR9006-2 on pharmacokinetics, safety, and tolerability when administered separately or co-administered to healthy male volunteers.

DETAILED DESCRIPTION:
A total of 36 subjects will be enrolled in one sequence group. The investigational products will be administered according to the treatment groups (T, M, T+M) assigned to one sequence group in Period 1, Period 2, and Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are given sufficient explanations about the trial objectives and contents as well as properties of investigational drugs before participating in the trial, and will voluntarily express their consent by signing an IRB-approved written consent to participate in the trial.
2. Healthy male adults aged 19 to 55 years at screening.
3. The subject's weight is 50kg or more and body mass index (BMI) is 18.0 or more but 30.0 or less.

Exclusion Criteria:

1. Those who have history of clinically significant diseases including hypersensitivity reaction, intolerability and anaphylaxis to major ingredients (Tamsulosin and Mirabegron) and other ingredients of investigational products, Food Yellow No. 5 (Sunset Yellow FCF) or Sulfonamide.
2. Those who have a history of clinically significant diseases related to liver, kidney, digestive system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hemato-oncology system, cardiovascular system (including orthostatic hypotension), etc.
3. Those who have medical history of gastrointestinal system diseases (for example: Crohn's disease, peptic ulcer disease, etc.) and operations that may influence the absorption of investigational drugs. (However, appendectomy, hernia operation, endoscopic polypectomy and hemorrhoids/anal fissure/anal fistula surgeries are excluded.)
4. Those with abnormal findings from the screening tests (medical interview, vital signs, electrocardiography, physical checkup, blood test, urinalysis, etc.) are judged to have clinical significance.
5. Those who are positive to HBsAg, HCV Ab, HIV Ab, VDRL tests at screening.
6. Those with any of the following results at screening:

   * AST or ALT > twice the upper limit of normal range
   * T. bilirubin > twice the upper limit of normal range
   * Estimated glomerular filtration rate (e-GFR) < 60 mL/min/1.73m2 (MDRD method used)
7. Those with systolic blood pressure > 150 mmHg or < 90 mmHg, or diastolic blood pressure > 95 mmHg or < 60 mmHg from vital signs at screening.
8. Those who took drugs (prescription drugs, OTC, herbal medicine or nutritional supplements (vitamins, etc.)) 2 weeks before screening. (However, those may participate in the trial if their safety and study results are considered to be unaffected according to the investigator's judgment.)
9. Those who have a drug abuse problem (especially centrally acting drugs including sleeping pills, centrally acting pain reliever, opiates or psychoactive drugs) or have a history of drug abuse.
10. Those who have a history of continuous alcohol intake exceeding 21 units/week (1unit=10g=12.5mL) within 6 months before screening.
11. Those who have smoked more than 10 cigarettes a day within 6 months before screening.
12. Those who have participated in other clinical trials and have been administered with other investigational drugs 180 days prior to the estimated administration date of this study's investigational drugs (However, is not applicable if the investigational drugs from other trials are not administered).
13. Those who have given whole blood 8 weeks before screening, who have given plasma/platelet 4 weeks before screening or who have not expressed their consent for blood-donation prohibition between the period from the first administration and 30 days after the final administration of the investigational drugs.
14. Those who have not expressed their consent for diet restrictions (grapefruit, caffeine in particular) that can influence absorption, distribution, metabolism and excretion of investigational drugs in the period between 3 days before the first administration and the last visit.
15. Those who have not expressed their consent for using contraceptive measures (for example: contraceptive administration and implant or intrauterine devices, sterilization (vasectomy, tubal ligation, etc.)) and barrier methods (combined use of spermicides and condom, contraceptive vaginal diaphragm, contraceptive sponge or cervical cap) that are allowed for clinical trials in the period between the first administration of the investigational drugs and the last visit.
16. Others who are judged to be ineligible to participate in the trial by the investigator.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables - Maximum (peak) steady-state plasma drug concentration during a dosage interval(Cmax,ss) of Part A and B | 0~26 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Tamsulosin vs. Tamsulosin + Mirabegron) and Part B (Mirabegron vs. Mirabegron + Tamsulosin).
Pharmacokinetic variables - Area under the plasma concentration-time curve from time zero to time t(AUCt) of Part A and B | 0~26 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Tamsulosin vs. Tamsulosin + Mirabegron) and Part B (Mirabegron vs. Mirabegron + Tamsulosin).

SECONDARY OUTCOMES:
Pharmacokinetic variables - Time to reach maximum (peak) plasma concentration following drug administration at steady state (Tmax,ss) of Part A and B | 0~26 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Tamsulosin vs. Tamsulosin + Mirabegron) and Part B (Mirabegron vs. Mirabegron + Tamsulosin).
Pharmacokinetic variables - Minimum steady-state plasma drug concentration during a dosage interval (Cmin,ss) of Part A and B | 0~26 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Tamsulosin vs. Tamsulosin + Mirabegron) and Part B (Mirabegron vs. Mirabegron + Tamsulosin).

CONTACTS AND LOCATIONS:
Overall Officials: An-Hye Kim, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea